CLINICAL TRIAL: NCT00739570
Title: The Effect of Manipulations of the Lumbar Spine on Six Different Outcome Measures.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec a Montréal (Other)
Responsible Party: Dr. Richard Roy, UQAM
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 071970
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Low Back Pain
Keywords: Activator; EMG; Thermography; Diagnostic; X-Rays
MeSH Terms: conditions — Low Back Pain; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention)
- 2 (Active Comparator): Activator chiropractic technique basic scan protocol
  Interventions: Device: AAI signature IV AMCT

INTERVENTIONS:
Device: AAI signature IV AMCT — Chiropractic adjustments of the lumbar spine following the activator basic scan protocol
  Other Names: Activator adjusting instrument signature series version IV
  Arms: 2

SUMMARY:
1. Evaluation of the effect of a chiropractic adjustment (Manually Assisted Mechanical Force)on
2. surface Static EMG
3. Paraspinal cutaneous temperature
4. Range of Motion
5. Dynamic EMG
6. Blood hormones (Interleukin-6 and C-Reactive protein)

DETAILED DESCRIPTION:
The chiropractic profession utilizes different outcome measures to evaluate and validate the chiropractic adjustments or the necessity for care. Some of these outcome measures have never been compared to each other under the same treatment and trials. In addition, blood analysis was added to measure the change in the inflammatory processes for the treatment period.

Outcome measures The outcome measures that we measured are: activities of daily living questionnaire (Oswestry disability index) , Interleukin-6 (IL-6), C-Reactive Protein (CRP), lateral bending x-ray analysis, heart rate variability (HRV), paraspinal temperature, paraspinal surface EMG (sEMG) static and dynamic (flexion, lateral bending and rotation) and the range of motion (ROM) in flexion and extension.

Activities of daily living questionnaire The modified Oswestry disability index 25 was utilized. It comprises ten questions that evaluate the capacity of the patient to function doing his daily activities and how the patient rates himself on a scale from A to F. The value of A= 0 and each subsequent letter as an ascending numerical value, B=1 to F=5. The maximum total for all ten questions is 50. The total for all the answers is tabulated and multiplied by two to give a percentage of dysfunction due to lumbar pain.

Blood Samples The blood samples were collected for Interleukin-6 (IL-6) and for C-Reactive Protein (CRP), by a trained nurse with a valid license for the province of Quebec. The IL-6 blood sample was collected in a lavender tube (4.0 ml, BD Vacutainer, K2 EDTA, lot 7344830, BD, Franklin Lakes, New Jersey, USA) and the sample was left at room temperature for 15 minutes then it was centrifuge for 15 minutes at 1000g, it was immediately decanted and the plasma was transferred via disposable transfer pipette ( Category number 13-711-7 Fisher Scientific, Pittsburgh, Pennsylvania, USA) into Eppendorf tubes (Sarstedt, Nümbrecth, Germany), the tube was closed and the tube was put on dry ice until it was delivered at the laboratory of the Hôpital St-Luc in Montréal. The CRP blood sample was collected in a yellow tube (5.0 ml, BD Vacutainer, SST, lot 8032322, BD, Franklin Lakes, New Jersey, USA) and the sample was left at room temperature for 15 minutes then it was centrifuge for 15 minutes at 1000g, it was immediately decanted and the serum was transferred via disposable transfer pipette ( Category number 13-711-7Fisher Scientific, Pittsburgh, Pennsylvania, USA) into Eppendorf tubes (Sarstedt, Nümbrecth, Germany), the tube was closed and the tube was put on dry ice until it was delivered at the laboratory of the Hôpital St-Luc in Montréal. All the needles were disposed after a single use in a biohazard container (BD, Sharps collector, reference number 305648, lot 7103001, BD Medical, Oakville, Ontario) provided by the Centre Local de Services de Santé (C.L.S.C.), an organism from the Quebec Ministry of Health. The analyses were performed at the laboratory of Hôpital St-Luc in Montreal under the supervision of Dr. Line Labrecque PhD in biochemistry. The results were provided by electronic means with the patient's code.

X-ray analysis The participants were x-rayed for the lumbar spine. AP lateral bending films in the left and right lateral bending position 27, 28, 29 were taken in the end position of the movement as the patient would stop once the end position was reached; the central ray was going through an area seven to eight centimeters above the top of the iliac crest. The lateral film was done with the central ray going through L-5. The radiographs were analyzed by two independent chiropractors, one chiropractor did the pre treatment analysis and the other chiropractor did the post analysis. The treating chiropractor was allowed to view the radiographs, for the purpose of treatment, after the initial analyses were terminated.

HRV measurement and analysis. A commercially available heart rate monitor (Suunto watch, model T6, FitzWright Company Ltd., Langley, BC, Canada) was used. The data recordings obtained from the heart rate monitor were analyzed for a five minute interval starting at the 80 Hz mark, in order to eliminate "bruit" from the initial positioning of the subject on the table, finishing at the 380 Hz mark,. The analysis was performed with a personal computer using custom software 15 (Kubios, Biosignal Analysis and Medical Imaging Group, Department of Physics, University of Kuopio, Kuopio, Finland) for several HRV parameters, as described below. As well, as mentioned above, there were no attempts to blind the assessment since the data were recorded directly into the heart rate monitor. Thus, the examiner could not know the value during measurement. The risk of influencing HRV was kept to a minimum by insuring that the interaction, between the subject and the examiner, limited itself to the installation and removal of the recording apparatus.

HRV Variables. The following variables were evaluated, mean R-R interval (Mean RR), the standard deviation between r-r intervals (SDNN), the number of pairs of adjacent NN intervals differing by more than 50 ms (NN 50 Count) and the proportion of NN intervals differing by more than 50 ms = NN50 divided by total number of NN intervals (pNN 50%), the very low frequency between (VLF); the normalized spectral components between 0 and 0.04 Hz , the low frequency (LF); similarly, the normalized spectral components between 0.04 and 0.15 Hz, the high frequency (HF); the normalized spectral power components were summed between 0.15 and 0.4 Hz and the ratio LF/HF 16. The HF band is related to the parasympathetic nervous system efferent activity 17 and is synchronized to respiratory rhythms 16. The LF band is related to both the sympathetic nervous system and parasympathetic nervous system efferent activity 18 and the cardiac sympathetic and parasympathetic nerve activity 16. The VLF band is not well defined but appears to be related to thermoregulation 16 renin-angiotensin-aldosterone systems 19-20, parasympathetic mechanisms 21, both the parasympathetic 21 and sympathetic branches of ANS affect VLF 22 and the humoral system 23, 24. The LF/HF ratio is used to indicate balance between the sympathetic nervous system and parasympathetic nervous system efferent tone 18. Thus, a change in this score might indicate either a parasympathetic nervous system or a sympathetic nervous system tonal change.

Myovision Instrumentation package The sEMG static and dynamic were connected to the Myovision 8000™ performance multi function sEMG (serial number 833830, Precision Biometrics Inc. 981-A Industrial Road San Carlos, California, USA. 94070). The thermal, ROM probes and the Myovision 8000™ were connected in the vision port 2 (serial number H002973, Precision Biometrics Inc. 981-A Industrial Road San Carlos, California, USA. 94070). The Vision port™ was connected to the computer via a USB connector.

ELIGIBILITY:
Inclusion Criteria:

Participants

* Written informed consent was obtained from all participants.

Control group

The inclusion criterion:

* All participants were receiving maintenance chiropractic care
* All participants would not have any treatment during the two week span of the research project
* All participants were examined and x-rayed and were evaluated for all the same outcome measures.

Treatment group:

* All participants were recruited via an announcement in the newspaper, Le Messager de LaSalle, during the period from July 6th to the 20th 2008.
* The participants were suffering from a chronic low back condition of at least three months in duration.
* All participants were examined and x-rayed and were evaluated for all the same outcome measures.

Exclusion Criteria:

* None

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index, Functional x-rays, Range of Motion, Static EMG, Dynamic EMG, Paraspinal cutaneous temperature, | August 2008

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Roy, DCMScPhD(c), Principal Investigator — Université du Québec a Montréal
Locations (1):
- Chiro-clinique Richard Roy, LaSalle, Quebec, Canada